CLINICAL TRIAL: NCT03491410
Title: Breast Cancer Active Surveillance Alternative Option, Can Aspirin Make the Difference?
Brief Title: Breast Cancer Active Surveillance, Alternative Option, Aspirin Included
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Hospitalar Lisboa Ocidental (Other Government)
Responsible Party: Principal Investigator, Zacharoula Sidiropoulou, Principal Investigator, Centro Hospitalar Lisboa Ocidental
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHLOBREASTASP
Record Dates: First submitted 2018-03-22; First posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: Metastatic; Active Surveillance
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 (Placebo Comparator): Arm 1: standard Unit´s protocol + placebo
  Interventions: Drug: Placebo Oral Tablet
- B (Experimental): Arm 2: standard Unit´s protocol + aspirin
  Interventions: Drug: Aspirin Low Dose

INTERVENTIONS:
Drug: Aspirin Low Dose — Low-Dose Aspirin is to be added in the standard patient´s treatment
  Arms: B
Drug: Placebo Oral Tablet — Placebo is to be added in the standard patient´s treatment
  Arms: 1

SUMMARY:
Experimental, clinical, and epidemiological studies have all demonstrated the strong association between chronic inflammation and cancer, and many studies have correlated the prolonged presence of the inflammatory milieu with an increased risk for developing cancer.(1) Although the potential mechanism for aspirin preventing breast cancer is not known, possible pathways may involve platelets, inflammation, cyclooxygenase (COX) 2, hormones, or PI3 kinase. (2).

In actual clinical practice there exist clear guidelines for the use of aspirin in colorectal cancer but no such guidelines exist for the use of aspirin in breast cancer patients.

In the Unit´s proper experience, in patients under active surveillance and metastatic ones some present very good responses both in the neoadjuvant and in the metastatic setting but investigators intend to provide evidence and not just the experience. This study patients are proposed to combine their standard treatment with aspirin.

DETAILED DESCRIPTION:
Breast cancer patients with diagnosis of Ductal or Lobular Invasive Carcinoma or CDis that refuse to underwent surgery or are not qualified for, and independently of age or of their actual staging, are going to be allocated, randomly and in double masked way to one of two arms:

Arm 1: standard Unit´s protocol + placebo Arm 2: standard Unit´s protocol + aspirin

ELIGIBILITY:
Inclusion Criteria:

Every adult (above 18) y.o.patient with histologic diagnosis of Breast Cancer that refuse or is not suitable for surgical treatment, or with metastatic disease, remaining this way in an "active surveillance"

Exclusion Criteria:

Allergy or toxicity to aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3 years
  Patients Overall survival in arm 2 superior to the arm 1

SECONDARY OUTCOMES:
Metastatic Disease Stability | 1 year
  Metastatic disease stability (non progression) determined by imaging (ecography, CT,PET-CT or Bone Scintigraphy) in arm 2 superior to the arm 1
Tumor response till patient decides to exit the active surveillance | 6 months
  Tumor response till patient decides to exit the active surveillance

CONTACTS AND LOCATIONS:
Overall Officials: Zacharoula Sidiropoulou, MD, Principal Investigator — Centro Hospitalar Lisboa Ocidental

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen WY, Holmes MD. Role of Aspirin in Breast Cancer Survival. Curr Oncol Rep. 2017 Jul;19(7):48. doi: 10.1007/s11912-017-0605-6. PMID 28597105
- [Result] Keibel A, Singh V, Sharma MC. Inflammation, microenvironment, and the immune system in cancer progression. Curr Pharm Des. 2009;15(17):1949-55. doi: 10.2174/138161209788453167. PMID 19519435